CLINICAL TRIAL: NCT05161780
Title: Evaluation of Endoscopic Surgical Field Clarity Using Hot Saline Versus Lactated Ringer's Irrigation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carl Snyderman (Other)
Responsible Party: Sponsor-Investigator, Carl Snyderman, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21110081
Record Dates: First submitted 2021-12-02; First posted 2021-12-17 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Irrigation
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will consist of 30 patients undergoing skull base surgery for a Pituitary Adenoma. This study will be a prospective double blinded randomized controlled trial examining the efficacy of normal saline versus Lactated Ringer's in achieving clarity of the surgical field during endoscopic skull base surgery.
Who Masked: Investigator
Masking Description: The surgeon will be blinded to the type of irrigation being used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline (Active Comparator): This study will be a prospective double blinded randomized controlled trial. Fifteen patients will be randomly assigned to the normal saline group using a random number generator.
  Interventions: Drug: Normal Saline
- Lactated Ringer's Irrigation (Experimental): This study will be a prospective double blinded randomized controlled trial. Fifteen patients will be randomly assigned to the lactated reinger group using a random number generator.
  Interventions: Drug: Lactated Ringer's Irrigation

INTERVENTIONS:
Drug: Lactated Ringer's Irrigation — Lactated Ringers at 40C will be used for the entirety of the surgery including the approach and exposure of the tumor as well as tumor resection, After surgery, two blinded skull base surgeon reviewers will rate the clarity of the endoscopic field of view at the recorded intervals. The surgical field will be graded using a widely accepted numeric integer (Boezaart) scale.
  Arms: Lactated Ringer's Irrigation
Drug: Normal Saline — Normal Saline at 40C will be used for the entirety of the surgery including the approach and exposure of the tumor as well as tumor resection, After surgery, two blinded skull base surgeon reviewers will rate the clarity of the endoscopic field of view at the recorded intervals. The surgical field will be graded using a widely accepted numeric integer (Boezaart) scale.
  Arms: Normal Saline

SUMMARY:
This study is designed to determine whether Normal Saline or Lactated Ringer's irrigation is superior in maintaining superior endoscopic surgical field clarity in surgery for pituitary adenoma.

DETAILED DESCRIPTION:
The aims of this study are to determine whether the endoscopic surgical view is objectively clearer using Normal Saline versus Lactated Ringer's Irrigation during endoscopic skull base surgery for pituitary adenoma. Other objectives include determining whether lactated Ringer's irrigation decreases total estimated blood loss and whether use of lactated Ringer's irrigation shortens surgical time.

Hot saline irrigation at 40 degrees Celcius has been shown to improve endoscopic surgical field clarity and its use is common practice in both endoscopic inflammatory sinus surgeries and skull base procedures. Saline irrigation dilutes blood in the surgical field keeping the endoscopic view clean and more bloodless and the elevated temperature promotes hemostasis.

Preliminary evidence suggests that the use of calcium-containing irrigant may further improve endoscopic surgical views. This mechanism is thought to be mediated through the activation of platelets and providing a calcium source to calcium-dependent factors in the coagulation cascade thereby promoting hemostasis. Using lactated Ringer's, a calcium-containing fluid, may result in improved surgeon visualization, decreased blood loss, and decreased complications during endoscopic approaches to the skull base.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a primary pituitary adenoma, macro or micro adenoma.

Exclusion Criteria:

* Age <18
* Pregnancy
* Revision surgery
* Non-surgical candidate due to medical, surgical, or anesthesia contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Boezaart scale rating video clips | 10 minutes
  Rating for each of the three recorded video clips per patient following tumor ablation. The Boezaart is an ordinal scale 0 = No bleeding 1 = Minimal bleeding: Not a surgical nuisance and no suction required 2 = Mild bleeding: Occasional suction required, but does not affect dissection 3 = Moderate bleeding: Slightly compromises surgical field, frequent suction required 4 = Severe bleeding: Significantly compromises surgical field, frequent suction required, bleeding threat field just after removal of suction 5 = Massive bleeding: Prevent dissection.
Boezaart scale rating video clips | 10 minutes
  rating for each of the three recorded video clips per patient after 10 minutes of irrigation. The Boezaart is an ordinal scale 0 = No bleeding 1 = Minimal bleeding: Not a surgical nuisance and no suction required 2 = Mild bleeding: Occasional suction required, but does not affect dissection 3 = Moderate bleeding: Slightly compromises surgical field, frequent suction required 4 = Severe bleeding: Significantly compromises surgical field, frequent suction required, bleeding threat field just after removal of suction 5 = Massive bleeding: Prevent dissection.
Boezaart scale rating video clips | 10 minutes
  rating for each of the three recorded video clips per patient at the completion of hemostasis. The Boezaart is an ordinal scale 0 = No bleeding 1 = Minimal bleeding: Not a surgical nuisance and no suction required 2 = Mild bleeding: Occasional suction required, but does not affect dissection 3 = Moderate bleeding: Slightly compromises surgical field, frequent suction required 4 = Severe bleeding: Significantly compromises surgical field, frequent suction required, bleeding threat field just after removal of suction 5 = Massive bleeding: Prevent dissection..
Time | 10 minutes
  Time between tumor ablation and the completion of hemostasis, or total irrigation time for patients undergoing normal saline or Lactated Ringer's irrigation during their surgical case.

SECONDARY OUTCOMES:
Estimated Blood Loss (EBL) | 15 min
  (EBL) per case and total operative time

CONTACTS AND LOCATIONS:
Overall Officials: Carl Snyderman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No